CLINICAL TRIAL: NCT01085838
Title: Phase I-II Trial of Erlotinib in Higher Risk Myelodysplastic Syndrome
Brief Title: Erlotinib in Higher Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-ERLOTINIB-08
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2013-03

CONDITIONS: Myelodysplastic Syndrome
Keywords: Erlotinib; myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): The first cohort of 5 patients will start with a dosage of 100 mg erlotinib daily
  Interventions: Drug: Erlotinib
- Cohort 2 (Experimental): The second cohort of patients will receive 150 mg of erlotinib daily
  Interventions: Drug: Erlotinib
- Cohort 3 (Experimental): The third cohort of five patients will be enrolled to receive 300 mg of erlotinib daily
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib oral capsule, 100, 150, or 300 mg/day during 12 weeks at study start
  Other Names: OSI-774

SUMMARY:
The aim of this study is to evaluate the toxicity and therapeutic efficacy of erlotinib in high-risk myelodysplastic syndrome (MDS) patients (with at least 10% of bone marrow blasts) ineligible for or having failed intensive chemotherapy and ineligible or after failure of treatment with a hypomethylating agent.

DETAILED DESCRIPTION:
This is a phase I-II multicenter, open label, sequential cohort dose escalation study of erlotinib designed to assess the safety and efficacy of a daily administration of erlotinib in high risk MDS patients.

Five patients per cohort will be enrolled into sequential cohorts receiving increasing dosages of erlotinib. The first cohort of 5 patients will start with a dosage of 100 mg erlotinib daily. Response will be determined after 12 weeks of treatment (or earlier upon major hematologic improvement, whichever event occurs first). At the completion of each cohort, defined as the fifth subject completing the week 12 visit, the safety review panel will be responsible for making the decision as to whether the next cohort will begin, an intermediate dose cohort will be added, or if additional subjects will be enrolled into an earlier dose cohort.

Upon agreement of the safety review panel, the second cohort of patients will receive 150 mg of erlotinib daily, and - upon agreement of the safety review panel - the third cohort of five patients will be enrolled to receive 300 mg of erlotinib daily.

Since it is to be expected that the therapeutically required dosage of erlotinib is higher than the dosage for which a patient was initially enrolled (i.e. patient enrolled in the first cohort receiving 100 mg daily), dosage of erlotinib should be increased (for the same patient) to the next higher level, if no response is documented after 12 weeks of continuous treatment and no grade III or IV toxicity is documented. In contrast, responders will continue their treatment with the same dosage of erlotinib until grade III or IV toxicity arises or treatment loses efficacy (as defined by relapse/progression of the disease).

Consequently, this study plans to enrol 15 patients in 3 cohorts of 5 patients. Once the dose limiting toxicity has been defined, additional confirmatory subjects (20) will be enrolled into the appropriate lower dose as recommended by the safety review panel.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MDS according to the WHO classification, but also including RAEB in transformation as defined by the FAB classification (that is patients with up to 30% of blasts in the bone marrow), with the exception of patients with preceding myeloproliferative syndrome or LMMC;
2. Higher-risk MDS as defined by a IPSS score >1 (IPSS: Int-2 or High);
3. Life expectancy > 3 months;
4. Percentage of bone marrow blasts >10 and below 30%;
5. Ineligible for or having failed intensive chemotherapy and ineligible for or having failed previous therapy with a hypomethylating agent;
6. Age ≥ 18 years;
7. Written informed consent;
8. Patient must understand and voluntarily sign consent form;
9. Patient must be able to adhere to the visit schedule as outlined in the study and follow protocol requirements;
10. ECOG performance status between 0-2 at the time of screening;
11. Females of childbearing potential (defined as a sexually mature woman who has not undergone a hysterectomy or who is not naturally postmenopausal for at least 24 consecutive months, that is who has had menses at any time during the preceding 24 consecutive months) have to have a negative pregnancy test;
12. Adequate contraceptive methods should be carried out by all patients during therapy and for at least 2 weeks after completing therapy.
13. No existing contra-indication to treatment with erlotinib.
14. Health insurance.

Exclusion Criteria:

1. Serum creatinine ≥ 1.5 x the upper limit of normal, or creatinine clearance ≤60 mL/min.
2. Concomitant treatment with NSAIDS, warfarin, omeprazole, ranitidine or inducers (i.e. rifampicin, phenytoin; carbamazepin) or inhibitors (i.e. ketoconazole, ciprofloxacin, clarithromycin, voriconazole) of CYP3A4;
3. Inadequate liver function as defined by a serum bilirubin ≥ 1.5 x the upper limit of normal (except in the case of confirmed moderate unconjugated hyperbilirubinemia due to intramedullary hemolysis, as observed frequently in MDS), and/or ASAT/ALAT/GGT levels ≥2 x the upper limit of normal;
4. Known HIV-positivity;
5. Any serious medical condition or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he or she participates in the study;
6. Vitamine B12 or folate deficiency;
7. Pregnant or lactating females;
8. Use of cytotoxic chemotherapeutic agents or experimental agents (agents that are not commercially available) for the treatment of MDS within the 28 days preceding study entry;
9. Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast), unless the subject has been disease-free for ≥3 years;
10. Patients with a history of corneal disorders or another active ophthalmic disorder, active infections or other concomitant serious and uncontrolled medical conditions.
11. History of interstitial lung disease or any active pulmonary disease.
12. Patients with a history of myeloproliferative syndrome or LMMC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to estimate the overall response rate (CR, PR, mCR The primary objective is to estimate the overall response rate (CR, PR, mCR and HI according to the IWG 2000 and 2006 criteria) in patients treated with erlotinib. | After 12 weeks treatment

SECONDARY OUTCOMES:
·assessment of response duration | While patient is on study/during follow-up.
· survival | While patient is on study/during follow-up.
· treatment-related toxicity; | While patient is on study/during follow-up.
· correlation of prognostic parameters, response and survival, with the assessed biological parameters; | While patient is on study/during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Thepot, MD, Principal Investigator — GFM/Hôpital Angers; Lionel Ades, MD, Principal Investigator — GFM/Hôpital Saint Louis
Locations (14):
- France (14):
  - CHU d'Angers, Angers
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier du Mans, Le Mans
  - CHRU Huriez, Lille
  - CHRU de Limoges, Limoges
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU Nantes, Nantes
  - CHU Caremeau, Nîmes
  - Hopital St Louis, Paris
  - Hopital Cochin, Paris
  - Hopital Purpan-Medecine interne, Toulouse
  - Hopital Purpan, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No